CLINICAL TRIAL: NCT07231289
Title: Effects of Soundscapes on the Mood States, Stress, and Anxiety in Individuals With Fibromyalgia Syndrome: A Randomized, Triple-Blind, Placebo-Controlled 4×4 Crossover Trial
Brief Title: Effect of Soundscapes on Emotional Distress in Fibromyalgia: a 4×4 Crossover Trial
Acronym: FMSounDistress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Mármol, Associate Professor, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIBROSOUNDS2025
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Fibromyalgia Syndrome
Keywords: Acoustic environment; Anxiety; Blank tape; Broadband noise; Chronic pain; Chronic primary pain; Clinical trial; Crossover; Emotional distress; Fibromyalgia; Mental health; Natural sound; Pink noise; Soundscape; Stress; Urban sound; White noise
MeSH Terms: conditions — Fibromyalgia; Anxiety Disorders; Chronic Pain; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study employs a randomized, triple-blind, placebo-controlled crossover design based on a 4×4 Williams Latin square. Each participant receives all four interventions in a randomized, balanced sequence across four periods, with one-week washout intervals separating each session to mitigate residual effects. The design ensures equal representation of each condition across periods and sequences (uniform within sequences and periods), controlling for first-order carryover effects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employs a triple-blind design: intervention administrator, outcome assessor, and data analyst will be fully blinded, while participants will remain unaware (masked, not blinded) of the study hypotheses. The intervention administrator will be blinded to the audio content being delivered, as stimuli will be labeled with non-descriptive codes by a separate investigator. The outcome assessor will not be involved in the intervention and will be blinded to group allocation. Participants will be instructed not to disclose any intervention-related information. Any potentially unblinding data that could reveal group allocation will be masked before it reaches the outcome assessor. The data analyst will receive fully de-identified datasets, with groups labeled only as "Group A/B/C/D"; unblinding will occur only after all analyses have been completed and verified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence NBPU (Other): Participants assigned to this sequence receive natural soundscape exposure in Week 1, broadband sound active control in Week 2, placebo control (blank tape) in Week 3, and urban soundscape exposure in Week 4. Each session lasts 20 minutes, with one-week washout intervals between sessions.
  Interventions: Other: Natural soundscape exposure; Other: Urban soundscape exposure; Other: Broadband sound active control; Other: Blank tape
- Sequence UPBN (Other): Participants assigned to this sequence receive urban soundscape exposure in Week 1, placebo control (blank tape) in Week 2, broadband sound active control in Week 3, and natural soundscape exposure in Week 4. Each session lasts 20 minutes, with one-week washout intervals between sessions.
  Interventions: Other: Natural soundscape exposure; Other: Urban soundscape exposure; Other: Broadband sound active control; Other: Blank tape
- Sequence BUNP (Other): Participants assigned to this sequence receive broadband sound active control in Week 1, urban soundscape exposure in Week 2, natural soundscape exposure in Week 3, and placebo control (blank tape) in Week 4. Each session lasts 20 minutes, with one-week washout intervals between sessions.
  Interventions: Other: Natural soundscape exposure; Other: Urban soundscape exposure; Other: Broadband sound active control; Other: Blank tape
- Sequence PNUB (Other): Participants assigned to this sequence receive placebo control (blank tape) in Week 1, natural soundscape exposure in Week 2, urban soundscape exposure in Week 3, and broadband sound active control in Week 4. Each session lasts 20 minutes, with one-week washout intervals between sessions.
  Interventions: Other: Natural soundscape exposure; Other: Urban soundscape exposure; Other: Broadband sound active control; Other: Blank tape

INTERVENTIONS:
Other: Natural soundscape exposure — Participants receive a standardized 20-minute auditory exposure to curated natural soundscapes via high-fidelity open-back reference headphones powered by a DAC/amplifier and corrected for frequency response using calibration software. Participants are randomly assigned a recording with 10-second fade-in/out effects and calibrated to between 45 and 55 dB (Leq,20min). The stereo recordings (320-kbps MP3, 48 kHz/24-bit) feature biophony (e.g., bird vocalizations) and geophony (e.g., rainfall), free of urban sounds and selected for ecological validity based on predefined criteria: (i) recognizable/context-specific sounds; (ii) culturally neutral; (iii) foreground presence and depth; (iv) no prolonged silence; (v) no technical artifacts. During exposure, they lie supine in a 60° Fowler's position on a therapy table, with sensory input minimized through auditory isolation and controlled ambient conditions. The session involves active listening under continuous researcher supervision.
  Other Names: Experimental intervention N
Other: Urban soundscape exposure — Participants receive a standardized 20-minute auditory exposure to curated urban soundscapes, using the same equipment and technical specifications as all other intervention conditions. Each participant is randomly assigned a recording that is calibrated between 60 and 70 dB (Leq,20min), with 10-sec fade-in/fadeouts. The recordings feature anthropophony (e.g., unintelligible background speech) and technophony (e.g., transportation-related sounds), free of natural sounds and selected for ecological validity based on the same predefined criteria as the natural soundscapes. To prevent semantic processing, participants are pre-screened and post-session reconfirmed to ensure they do not understand the languages used. During exposure, participants lie supine in a 60° Fowler's position on a therapy table, with sensory input minimized through auditory isolation and controlled ambient conditions. The session involves active listening and is conducted under continuous researcher supervision.
  Other Names: Experimental intervention U
Other: Broadband sound active control — Participants receive a standardized 20-minute auditory exposure to broadband sounds (i.e., white or pink noise), using the same equipment and technical specifications as all other intervention conditions. Each participant is randomly assigned to one of the two noise types, with equal distribution across conditions. The stimuli are generated using professional audio software and calibrated to 50 dB (Leq,20min). During exposure, participants lie supine in a 60° Fowler's position on a therapy table, with sensory input minimized through auditory isolation and controlled ambient conditions. The session involves active listening and is conducted under continuous researcher supervision.
  Other Names: Active control
Other: Blank tape — Participants receive a standardized 20-minute exposure to blank audio (silence), using the same equipment and technical specifications as all other intervention conditions. At study onset, participants are informed they will hear a range of environmental sounds, including some that may be inaudible (i.e., present but beyond the range of human hearing). During the placebo condition, a blank recording is played, producing silence, while participants remain unaware of whether they are receiving an active or placebo stimulus. This attention-control condition ensures procedural consistency while delivering no auditory stimulation. During exposure, participants lie supine in a 60° Fowler's position on a therapy table, with sensory input minimized through auditory isolation and controlled ambient conditions. The session involves active listening and is conducted under continuous researcher supervision.
  Other Names: Placebo attention control

SUMMARY:
This study tests whether different types of sounds can help reduce emotional distress in people with fibromyalgia. Fibromyalgia is a condition that causes widespread muscle and joint pain and makes people extra sensitive to sounds and other sensations. Many people with fibromyalgia also struggle with emotional distress symptoms. About half of people with fibromyalgia (54 out of 100) have depression symptoms, while 55 out of 100 also have anxiety symptoms.

Researchers want to know if listening to environmental sounds can help people with fibromyalgia feel less distressed. The study will include four different types of sounds:

* Natural sounds (like birds singing, water flowing, and wind in trees)
* City sounds (like traffic, people talking, machines)
* Broadband sounds (steady sounds like white noise)
* Silence (no sound at all)

People with fibromyalgia who are between 18 and 64 years old may be able to join. The study takes 4 weeks total. Each person will visit the research center 4 times over these weeks. Each visit takes about 1 hour. Visits are scheduled 1 week apart. During each visit, participants will:

1. Answer questions about how they feel before listening to sounds.
2. Lie comfortably and listen to one type of sound for 20 minutes through headphones.
3. Answer the same questions again after listening.

Each person will try all 4 types of sounds in a random order. This helps researchers compare how each sound affects the same person.

Before and after each sound session, participants will fill out questionnaires about:

* Their mood states at the moment of evaluation
* How stressed they feel at the moment of evaluation
* How anxious they feel at the moment of evaluation

These questionnaires have been tested in many studies and work well for people with chronic pain conditions.

Participants' mood, stress, and anxiety levels might change after listening to certain sounds. If the study shows that sounds help, this could lead to new treatment options and preventive measures that are easy to use and would be safe and cost much less than medications.

DETAILED DESCRIPTION:
This study investigates whether distinct soundscapes can alleviate emotional distress symptoms in individuals with fibromyalgia syndrome. The study's theoretical foundation is grounded in converging evidence from environmental neuroscience and psychology research demonstrating that auditory stimuli can significantly influence emotional processing through neural pathways connecting the auditory cortex with brain areas involved in emotional regulation. By investigating how different soundscapes influence emotional distress, this research may contribute to the field of environmental psychology, as well as inform environmental health policies and acoustic design strategies for healthcare settings.

Soundscapes represent acoustic environments that are perceived, experienced, and interpreted within specific contexts. For research purposes, soundscapes are categorized based on their sources: natural soundscapes comprise biophonies (sounds produced by non-human living organisms) and geophonies (sounds generated by non-biological natural processes), while urban soundscapes feature anthropophonies (human-generated sounds) and technophonies (sounds produced by mechanical and technological sources).

Emerging neuroscientific research has identified direct neural pathways between the auditory cortex and emotion-processing brain areas, including the limbic and paralimbic regions. These auditory-emotion connections may provide a neurobiological foundation for investigating how environmental soundscapes might modulate emotional states in populations with altered sensory processing. Moreover, numerous studies conducted in healthy populations suggest that soundscapes can influence mood states and stress levels. Natural soundscapes have been shown to elicit distinct neural signatures compared to urban soundscapes, with differential effects on emotional distress symptoms.

Fibromyalgia syndrome affects approximately 2 to 3% of the global population and is commonly associated with emotional distress, with clinical symptoms of depression and anxiety occurring in 54% and 55% of affected individuals, respectively. This high prevalence of emotional comorbidity significantly impacts various aspects of life in this population. The hypothalamic-pituitary-adrenal axis dysfunction observed in fibromyalgia may contribute to altered stress responsivity and emotional regulation difficulties. Furthermore, the chronic pain experience itself can precipitate and maintain emotional distress through various psychological mechanisms. The substantial emotional burden associated with fibromyalgia necessitates efficacious strategies that can address emotional distress symptoms characteristic of this condition.

The use of environmental acoustic stimuli to influence emotional distress symptoms may offer a promising management strategy in individuals with fibromyalgia. This proposition is supported by two core characteristics of the condition. First, fibromyalgia is associated with increased sensory sensitivity, which may heighten responsiveness to acoustic features of the environment. Second, emotion regulation difficulties have been identified as a key factor mediating the relationship between fibromyalgia symptoms and emotional distress. In particular, individuals with fibromyalgia often demonstrate reduced efficacy in employing adaptive emotion regulation strategies, such as cognitive reappraisal and emotional acceptance. These limitations may contribute to the persistence and intensification of affective symptoms. Together, these factors indicate that environmental sounds capable of modulating emotional distress symptoms through non-cognitive mechanisms represent a theoretically grounded and clinically relevant intervention approach for this population.

The general objective (GO) of this study is to:

GO1. Investigate whether exposure to distinct soundscapes differentially modulates emotional distress variables in individuals with fibromyalgia syndrome.

The specific objectives (SO) are to:

SO1. Compare the effects of natural and urban soundscapes with those of broadband sound (active comparator) and silence (attention-placebo control) on mood states, perceived stress, and state anxiety.

SO2. Determine the relative efficacy of natural versus urban soundscapes in modulating mood states, perceived stress, and state anxiety.

SO3. Quantify and characterize the magnitude and direction of within-group pre-post changes in mood states, perceived stress, and state anxiety following exposure to natural and urban soundscapes.

The primary hypothesis (PH) is:

PH1. Exposures to distinct soundscape categories will differentially modulate total mood disturbance in individuals with fibromyalgia syndrome, with the following specific contrasts:

PH1.1. Natural soundscape exposure will result in lower total mood disturbance compared to the attention-placebo control (silence).

PH1.2. Natural soundscape exposure will result in lower total mood disturbance compared to broadband sound active control.

PH1.3. Urban soundscape exposure will result in higher total mood disturbance compared to the attention-placebo control.

PH1.4. Urban soundscape exposure will result in higher total mood disturbance compared to broadband sound active control.

PH1.5. Natural soundscape exposure will result in lower total mood disturbance compared to urban soundscape exposure.

The secondary hypotheses (SH) are:

SH1. Exposures to distinct soundscape categories will differentially modulate perceived stress and state anxiety in individuals with fibromyalgia syndrome, with the following specific contrasts:

SH1.1. Natural soundscape exposure will result in lower perceived stress and state anxiety compared to the attention-placebo control.

SH1.2. Natural soundscape exposure will result in lower perceived stress and state anxiety compared to broadband sound active control.

SH1.3. Urban soundscape exposure will result in higher perceived stress and state anxiety compared to the attention-placebo control.

SH1.4. Urban soundscape exposure will result in higher perceived stress and state anxiety compared to broadband sound active control.

SH1.5. Natural soundscape exposure will result in lower perceived stress and state anxiety compared to urban soundscape exposure.

SH2. Exposure to natural soundscapes will produce a significant pre-post reduction in total mood disturbance, perceived stress, and state anxiety.

SH3. Exposure to urban soundscapes will produce a significant pre-post increase in total mood disturbance, perceived stress, and state anxiety.

The study design optimizes statistical efficiency by allowing within-subject comparisons while controlling period effects. The auditory exposure sessions are conducted in a controlled laboratory environment, maintaining a consistent room temperature and relative humidity.

An a priori power analysis was conducted using Monte Carlo simulations in R with the simr package. The sample size estimation was based on a linear mixed-effects model, with power evaluated via a likelihood ratio test. Model parameters were defined to detect a partial eta-squared of 0.075 with a two-tailed alpha level of 0.05, derived from literature on the impact of environmental sounds on total mood disturbance. The simulation assumed a total standard deviation of 25 for the primary outcome and an intra-class correlation of 0.5. To test the overall main effect of "treatment," a total of 56 participants provides 83.48% power (95% CI [82.42%, 84.50%]) based on 5000 simulations. To account for a potential attrition rate of 20%-including potential dropout, loss to follow-up, clinical reasons, and operational challenges-a total of 70 participants is required. To ensure balanced allocation across the four experimental sequences using a multiple of four, a final sample of 72 participants will be recruited.

The assessment protocol incorporates validated instruments specifically selected for their psychometric properties in chronic pain populations. It follows International Association for the Study of Pain consensus guidelines and incorporates core outcome domains recommended for chronic pain trials.

The primary and secondary analyses will employ linear mixed-effects models. The dependent variable will be defined as post-intervention outcome adjusted for baseline. Fixed effects will include treatment, sequence, period, and the treatment × period interaction term to assess potential carryover effects. Participants will be modeled as a random effect. If no statistically significant carry-over effect is detected at the 25% significance level, the interaction term will be excluded, and a reduced model will subsequently be re-estimated. The inferences will be based on the main effects from the final model. Following a significant omnibus F-test for the treatment effect, pairwise comparisons between interventions will be conducted using estimated marginal means with Bonferroni adjustment. As a sensitivity analysis, the prespecified covariate will be incorporated into the final model to assess its potential influence on the estimated treatment effects. Post-hoc analyses will include within-group changes from baseline, conducted using paired t-tests or Wilcoxon signed-rank tests, depending on the data's distributional properties. All hypothesis testing will be two-sided with an overall Type I error rate of 5%, and all analyses will adhere to the intention-to-treat (ITT) principle.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of fibromyalgia syndrome, documented in the medical record provided by the participant prior to enrollment.
* Normal hearing confirmed by a hearing test, defined as a mean threshold of ≤ 20 dB HL at 0.125, 0.25, 0.5, 1, 2, 4, 6, and 8 kHz.
* Ability to communicate in Spanish.
* Provision of signed written informed consent to participate in the research.

Exclusion Criteria:

* A diagnosis of misophonia or auditory processing disorders, as documented in the participant's medical record.
* Severe cognitive impairment, defined as a Mini-Mental State Examination score ≤ 17.
* Severe psychiatric disorders in the symptomatic phase.
* History of substance abuse in the past 12 months or current substance use disorder as reported by the participant.
* Changes in ongoing therapy during or within one month prior to study enrollment per participant self-reports.
* Any other serious or unstable medical condition that could interfere with study participation.
* Known allergies or hypersensitivity to study materials.
* Pregnancy, lactation, or being within three months postpartum at the time of study enrollment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-02-06 (Actual); Study Completion 2026-02-06 (Actual)

PRIMARY OUTCOMES:
Mood states | Change from immediately before to immediately after each 20-minute intervention session during each of the four crossover periods
  The positive and negative mood states will be assessed using the shortened version of the Profile of Mood States. This version comprises 30 self-administered items, evenly distributed across six mood dimensions: tension, depression, anger, fatigue, vigor, and friendliness. Each item is rated on a five-point Likert scale ranging from zero ("not at all") to four ("extremely"), yielding subscale scores ranging from zero to 20. Higher scores on the vigor and friendliness subscales reflect a more positive mood, whereas higher scores on the remaining subscales indicate greater negative mood. A total mood disturbance index is calculated by subtracting the sum of the positive mood subscales from the sum of the negative mood subscales. The total mood disturbance score ranges from -40 to 80, with lower scores denoting less mood disturbance-that is, a more positive overall mood.

SECONDARY OUTCOMES:
Perceived stress | Change from immediately before to immediately after each 20-minute intervention session during each of the four crossover periods
  Momentary psychological stress will be assessed using a 100-mm Visual Analog Scale. Participants will be presented with the following instruction: "Indicate how stressed you feel at the moment on the following ruler." The scale is anchored on the left by "none" and on the right by "as bad as it could be." The participant's response is recorded as the distance in millimeters from the left endpoint to their mark on the scale, yielding a single quantitative variable representing perceived stress. Lower scores indicate lower levels of perceived stress at the moment.
State anxiety | Change from immediately before to immediately after each 20-minute intervention session during each of the four crossover periods
  State anxiety will be assessed using a 100-mm Visual Analog Scale. Participants will be instructed as follows: "Please mark the line below with a vertical stroke to indicate how anxious you feel at the moment." The endpoints are labeled as "not at all anxious" and "extremely anxious" from left to right, respectively. The state anxiety score is determined by measuring the distance in millimeters from the far-left end to the participant's mark. Lower scores indicate lower levels of anxiety at the time of assessment.

OTHER OUTCOMES:
Connectedness to nature | Assessed immediately after the final 20-minute intervention session, following completion of all other outcome assessments during the fourth crossover period (Week 4)
  The Connectedness to Nature Scale assesses participants' attitudes toward nature. The self-report scale comprises 13 items rated on a five-point Likert scale, ranging from one ("strongly disagree") to five ("strongly agree"). The total score ranges from 13 to 65, with higher scores reflecting a greater sense of connectedness to nature.

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel Pérez Mármol, PhD, Principal Investigator — Department of Physiotherapy, Faculty of Health Sciences, University of Granada
Locations (1):
- Faculty of Health Sciences, University of Granada, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided